CLINICAL TRIAL: NCT01424553
Title: Respiratory Outcome at Adolescence of Very Low Birthweight Infants : the EPIPAGE Cohort
Brief Title: Respiratory Outcome at Adolescence of Very Low Birthweight Infants
Acronym: EPIPAGEADO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P100117
Record Dates: First submitted 2011-08-22; First posted 2011-08-29 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Premature Baby 26 to 32 Weeks; Bronchopulmonary Dysplasia
Keywords: Low birthweight; Bronchopulmonary dysplasia; Lung development; Airway obstruction; Asthma
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Airway Obstruction; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort (Other): All patients
  Interventions: Other: Prevention and follow-up of the patients pulmonary parameters

INTERVENTIONS:
Other: Prevention and follow-up of the patients pulmonary parameters — Respiratory symptoms and lung function will be evaluated in very low birth weight and term infants, born in 1997 and included in the French EPIPAGE cohort.
  Other Names: Prevention and follow-up pulmonary parameters

SUMMARY:
EPIPAGEADO is an observational study. Respiratory symptoms and lung function will be evaluated in very low birth weight and term infants, born in 1997 and included in the French EPIPAGE cohort.

DETAILED DESCRIPTION:
EPIPAGEADO is a multicenter observational study:- to evaluate respiratory symptoms and lung function at adolescence in very low birthweight (VLBW) children, to identify perinatal risk factors for persistent symptoms or impaired lung function tests at adolescence, to assess the exercise tolerance in VLBW children and to search for genetic susceptibility markers associated to impaired lung function.

The main criteria for analysis will be the forced expiratory volume in one seconde (FEV1) The study duration will be 36 months the number of centers will be 4 centers in France (Paris-Necker, Nantes, Lille, Rouen) The number of patients to be included will be 400, including 260 VLBW children without BPD, 40 VLBW children with BPD, 100 control children with birth at term.

ELIGIBILITY:
Inclusion criteria :

* Children born in 1997, and included at birth in the French EPIPAGE cohort
* Absence of severe neurologic impairment, with impossibility of reliable lung function tests
* Acceptance of the child and his/her parents

Exclusion criteria :

* Severe neurologic impairment, with impossibility of reliable lung function tests
* Absence of child's or parents' acceptance

Ages: 14 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 355 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume | Day 0 (at 14 - 15 years old)
  Forced expiratory volume in one seconde (FEV1) at 14-15 years

SECONDARY OUTCOMES:
Pulmonary parameters | Day 0 (at 14 - 15 years old)
  Pulmonary parameters will be assess by the measure of Vital capacity, total lung capacity, functional residual capacity, forced expiratory flow 25-75%, diffusing capacity for carbon monoxide, diffusing capacity for nitric monoxide, exhaled nitric monoxide, maximal oxygen consumption at exercise.
Standardized questionnaire for respiratory symptoms | Day 0 (at 14-15 years old)
Candidate-gene analysis, with SNPs known to be associated to bronchopulmonary dysplasia (BPD) | Day 0 (at 14-15 years old)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Delacourt, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Necker, Paris, France

REFERENCES:
- [Background] Hadchouel A, Marchand-Martin L, Franco-Montoya ML, Peaudecerf L, Ancel PY, Delacourt C; EPIPAGEADO study group. Salivary Telomere Length and Lung Function in Adolescents Born Very Preterm: A Prospective Multicenter Study. PLoS One. 2015 Sep 10;10(9):e0136123. doi: 10.1371/journal.pone.0136123. eCollection 2015. PMID 26355460
- [Background] Hadchouel A, Rousseau J, Roze JC, Arnaud C, Bellino A, Couderc L, Marret S, Mittaine M, Pinquier D, Verstraete M, Ancel PY, Delacourt C; EPIPAGEADO study group. Association between asthma and lung function in adolescents born very preterm: results of the EPIPAGE cohort study. Thorax. 2018 Dec;73(12):1174-1176. doi: 10.1136/thoraxjnl-2017-211115. Epub 2018 Mar 31. PMID 29605813
- [Background] Drummond D, Hadchouel A, Torchin H, Roze JC, Arnaud C, Bellino A, Couderc L, Marret S, Mittaine M, Pinquier D, Vestraete M, Rousseau J, Ancel PY, Delacourt C; EPIPAGEADO study group. Educational and health outcomes associated with bronchopulmonary dysplasia in 15-year-olds born preterm. PLoS One. 2019 Sep 11;14(9):e0222286. doi: 10.1371/journal.pone.0222286. eCollection 2019. PMID 31509594
- [Background] Drummond D, Hadchouel A, Le Bourgeois M, Roze JC, Marret S, Rousseau J, Ancel PY, Delacourt C. Decreased pulmonary capillary volume in adolescents born very preterm. Acta Paediatr. 2020 Mar;109(3):621-622. doi: 10.1111/apa.15023. Epub 2019 Oct 2. No abstract available. PMID 31531873